CLINICAL TRIAL: NCT01611818
Title: Low Intensity Versus Self-guided Internet-delivered Psychotherapy for Major Depression: a Multicenter, Controlled, Randomised Study
Brief Title: Low Intensity Versus Self-guided Internet-delivered Psychotherapy for Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier Garcia Campayo (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Javier Garcia Campayo, Principal Investigator, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI10/01083
Record Dates: First submitted 2012-05-23; First posted 2012-06-05 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Depression
Keywords: Depression; Computer-delivered psychotherapy; Randomized-controlled trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low intensity Internet-delivered psychotherapy (Other): Low intensity Internet-delivered psychotherapy + improved treatment as usual by GP.
  Interventions: Other: Low Intensity Internet-delivered psychotherapy
- Self-guided Internet-delivered psychotherapy (Other): Self-guided Internet-delivered psychotherapy + improved treatment as usual
  Interventions: Other: Self-guided Internet delivered psychotherapy
- Improved treatment as usual by GP (Other)
  Interventions: Other: Improved treatment as usual

INTERVENTIONS:
Other: Low Intensity Internet-delivered psychotherapy — Patients will be contacted by a researcher trained in psychotherapy. Patients can ask for questions or advice to psychotherapists during the study
  Arms: Low intensity Internet-delivered psychotherapy
Other: Self-guided Internet delivered psychotherapy — No contact with the therapists over the treatment period will be done.
  Arms: Self-guided Internet-delivered psychotherapy
Other: Improved treatment as usual — Any kind of treatment administered by the GP to the patient with depression
  Arms: Improved treatment as usual by GP

SUMMARY:
BACKGROUND: Major depression will become the second most important cause of disability in 2020. Computerised cognitive-behaviour therapy could be an efficacious and cost-effective option for its treatment. No studies on cost-effectiveness of low intensity vs self-guided psychotherapy have been carried out.

AIM: To assess the efficacy of low intensity vs self-guided psychotherapy for major depression in the Spanish health system.

METHODS: The study is made up of 3 phases: 1.- Development of a computerised cognitive-behaviour therapy for depression tailored to Spanish health system. 2.- Multicenter controlled, randomized study: A sample (N=450 patients) with mild/moderate depression recruited in primary care. They should have internet availability at home, not receive any previous psychological treatment, and not suffer from any other severe somatic or psychological disorder. They will be allocated to one of 3 treatments: a) Low intensity Internet-delivered psychotherapy + improved treatment as usual (ITAU) by GP, b) Self-guided Internet-delivered psychotherapy + ITAU or c) ITAU. Patients will be diagnosed with MINI psychiatric interview. Main outcome variable will be Beck Depression Inventory. It will be also administered EuroQol 5D (quality of life) and Client Service Receipt Inventory (consume of health and social services). Patients will be assessed at baseline, 3 and 12 months. An intention to treat and a per protocol analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression. It will be carried out with MINI International Neuropsychiatric Interview + scoring of moderate or mild depression using Beck Depression Inventory II. Cut-off point for this questionnaire is: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression [34, 35].
* Aged 18-65 years
* Able to understand and read Spanish
* Moderate or mild major depression
* Duration of symptoms longer than 2 weeks
* Access to Internet at home and having an email address.

Exclusion Criteria:

* Any psychological treatment during last year
* Severe psychiatric disorder in Axis I (alcohol/substances abuse or dependence, psychotic disorders or dementia)patients with severe depression (indicated by a Beck-II score of 29 or higher) who will be advised to consult their GP Receiving pharmacological treatment with antidepressants is not an exclusion criteria meanwhile, during the study period, treatment will not be modified or increased (decrease of pharmacological treatment is accepted).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Severity of depressive symptomatology measured by Beck Depression Inventory II | At baseline
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. This questionnaire has been used because it is recommended to assess depression in primary care patients in which comorbidity with medical disorders is frequent. The Spanish validated version of the questionnaire will be used.
Severity of depressive symptomatology measured by Beck Depression Inventory II | After the Internet-delivered psychotherapy program has been finished. We estimate 3 months on average to complete the program.
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. This questionnaire has been used because it is recommended to assess depression in primary care patients in which comorbidity with medical disorders is frequent. The Spanish validated version of the questionnaire will be used.
Severity of depressive symptomatology measured by Beck Depression Inventory II | 3 months after completing the psychotherapy program
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. This questionnaire has been used because it is recommended to assess depression in primary care patients in which comorbidity with medical disorders is frequent. The Spanish validated version of the questionnaire will be used.
Severity of depressive symptomatology measured by Beck Depression Inventory II | 12 months after completing the psychotherapy program
  This is one of the most widely questionnaires used to evaluate severity of depression in pharmacological and psychotherapy trials. This questionnaire has been used because it is recommended to assess depression in primary care patients in which comorbidity with medical disorders is frequent. The Spanish validated version of the questionnaire will be used.

SECONDARY OUTCOMES:
Socio-demographic variables. | At Baseline
  The following socio-demographic data will be collected: gender, age, marital status (single, married/relationship, separated/divorced, and widowed), education (years of education), occupation, economical level (in relation with Spanish minimum monthly salary that at the moment of the study was 640€).
Mini-International Neuropsychiatric Interview (MINI). | At Baseline
  This is a short structured diagnostic psychiatric interview that yields key DSM-IV and ICD-10 diagnoses. MINI can be administered in a short period of time and clinical interviewers need only a brief training. The MINI has been translated and validated in Spanish.
EuroQoL-5D questionnaire (EQ-5D - Spanish version) | At Baseline
  Generic instrument of health-related quality of life. It has two parts: part 1 records self-reported problems in each of five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is divided into three levels of severity corresponding to no problems, some problems, and extreme problems. Values range from 1 (best health state) to 0 (death). Part 2 records the subject's self-assessed health on a VAS, a 10 cm vertical line on which the best and worst imaginable health states score 100 and 0, respectively.
Client Service Receipt Inventory - adapted (CSRI - Spanish version) | At baseline
  Questionnaire for collecting information about use of healthcare and social care services and other economic impacts (such as time off work due to illness). The variant used in this study was designed to collect retrospective data on service utilization during the previous months after the last assessment. Data on baseline assess the previous three months before inclusion.
Overall Depression Severity and Impairment Scale | At baseline
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as level of avoidance, work/ school/home interference, and social interference associated with anxiety. The instructions orient the respondent to considerate wide range of anxiety symptoms (e.g., panic attacks, worries, flashbacks) when answering the questions, and the time frame is "over the past week". Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score.
Positive and Negative Affect Scale (PANAS) | At Baseline
  PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is 10 to 50. The instrument's psychometric properties are quite satisfactory. It has a validated Spanish version.
Credibility/expectancy questionnaire | At Baseline
  It is a quick and easy-to-administer scale for assessing treatment expectancy and rationale credibility. Credibility has been defined as how believable, convincing, and logical the treatment is, whereas expectancy refers to improvements that clients believe will be achieved. The aspects that address these two scales relate to: 1) treatment rationale, 2) treatment satisfaction, 3) degree to which I would recommend to a friend who had the same problem, 4) extent to which is considered to be useful in the same case, 6) extent to which the intervention would be considered aversive.
EuroQoL-5D questionnaire (EQ-5D - Spanish version) | After the Internet-delivered psychotherapy program has been finished. We estimate 3 months on average to complete the program.
  Generic instrument of health-related quality of life. It has two parts: part 1 records self-reported problems in each of five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is divided into three levels of severity corresponding to no problems, some problems, and extreme problems. Values range from 1 (best health state) to 0 (death). Part 2 records the subject's self-assessed health on a VAS, a 10 cm vertical line on which the best and worst imaginable health states score 100 and 0, respectively.
EuroQoL-5D questionnaire (EQ-5D - Spanish version) | 3 months after completing the psychotherapy program
  Generic instrument of health-related quality of life. It has two parts: part 1 records self-reported problems in each of five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is divided into three levels of severity corresponding to no problems, some problems, and extreme problems. Values range from 1 (best health state) to 0 (death). Part 2 records the subject's self-assessed health on a VAS, a 10 cm vertical line on which the best and worst imaginable health states score 100 and 0, respectively.
EuroQoL-5D questionnaire (EQ-5D - Spanish version) | 12 months after completing the psychotherapy program
  Generic instrument of health-related quality of life. It has two parts: part 1 records self-reported problems in each of five domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each domain is divided into three levels of severity corresponding to no problems, some problems, and extreme problems. Values range from 1 (best health state) to 0 (death). Part 2 records the subject's self-assessed health on a VAS, a 10 cm vertical line on which the best and worst imaginable health states score 100 and 0, respectively.
Client Service Receipt Inventory - adapted (CSRI - Spanish version) | After the Internet-delivered psychotherapy program has been finished. We estimate 3 months on average to complete the program
  Questionnaire for collecting information about use of healthcare and social care services and other economic impacts (such as time off work due to illness). The variant used in this study was designed to collect retrospective data on service utilization during the previous months after the last assessment. Data on baseline assess the previous three months before inclusion.
Client Service Receipt Inventory - adapted (CSRI - Spanish version) | 3 months after completing the psychotherapy program
  Questionnaire for collecting information about use of healthcare and social care services and other economic impacts (such as time off work due to illness). The variant used in this study was designed to collect retrospective data on service utilization during the previous months after the last assessment. Data on baseline assess the previous three months before inclusion.
Client Service Receipt Inventory - adapted (CSRI - Spanish version) | 12 months after completing the psychotherapy program
  Questionnaire for collecting information about use of healthcare and social care services and other economic impacts (such as time off work due to illness). The variant used in this study was designed to collect retrospective data on service utilization during the previous months after the last assessment. Data on baseline assess the previous three months before inclusion.
Overall Depression Severity and Impairment Scale | After the Internet-delivered psychotherapy program has been finished. We estimate 3 months on average to complete the program.
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as level of avoidance, work/ school/home interference, and social interference associated with anxiety. The instructions orient the respondent to considerate wide range of anxiety symptoms (e.g., panic attacks, worries, flashbacks) when answering the questions, and the time frame is "over the past week". Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score.
Overall Depression Severity and Impairment Scale | 3 months after completing the psychotherapy program
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as level of avoidance, work/ school/home interference, and social interference associated with anxiety. The instructions orient the respondent to considerate wide range of anxiety symptoms (e.g., panic attacks, worries, flashbacks) when answering the questions, and the time frame is "over the past week". Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score.
Overall Depression Severity and Impairment Scale | 12 months after completing the psychotherapy program
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as level of avoidance, work/ school/home interference, and social interference associated with anxiety. The instructions orient the respondent to considerate wide range of anxiety symptoms (e.g., panic attacks, worries, flashbacks) when answering the questions, and the time frame is "over the past week". Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score.
Positive and Negative Affect Scale (PANAS) | After the Internet-delivered psychotherapy program has been finished. We estimate 3 months on average to complete the program.
  PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is 10 to 50. The instrument's psychometric properties are quite satisfactory. It has a validated Spanish version.
Positive and Negative Affect Scale (PANAS) | 3 months after completing the psychotherapy program
  PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is 10 to 50. The instrument's psychometric properties are quite satisfactory. It has a validated Spanish version.
Positive and Negative Affect Scale (PANAS) | 12 months after completing the psychotherapy program
  PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is 10 to 50. The instrument's psychometric properties are quite satisfactory. It has a validated Spanish version.

CONTACTS AND LOCATIONS:
Overall Officials: Javier García Campayo, PhD, Principal Investigator — Miguel Servet Hospital & University of Zaragoza, Spain
Locations (6):
- Spain (6):
  - Hospital Parc Sanitari Sant Joan de Deu, Sant Boi de Llobregat, Barcelona
  - Health Science Research Institute, University Balearic Islands, Palma de Mallorca, Mallorca
  - Psychiatric Service. Hospital Vall D'Hebrón, Barcelona
  - Psychiatric Service. University Hospital Carlos Haya, Málaga
  - Valencia University and CIBER Physiopathology of Obesity and Nutrition. Carlos III Health Institute, Valencia
  - Department of Psychiatry. Miguel Servet University Hospital, Zaragoza

REFERENCES:
- [Background] Fernandez A, Saameno JA, Pinto-Meza A, Luciano JV, Autonell J, Palao D, Salvador-Carulla L, Campayo JG, Haro JM, Serrano A; DASMAP investigators. Burden of chronic physical conditions and mental disorders in primary care. Br J Psychiatry. 2010 Apr;196(4):302-9. doi: 10.1192/bjp.bp.109.074211. PMID 20357307
- [Background] Cuijpers P, van Straten A, van Oppen P, Andersson G. Are psychological and pharmacologic interventions equally effective in the treatment of adult depressive disorders? A meta-analysis of comparative studies. J Clin Psychiatry. 2008 Nov;69(11):1675-85; quiz 1839-41. doi: 10.4088/jcp.v69n1102. Epub 2008 Aug 12. PMID 18945396
- [Background] Andrews G, Issakidis C, Sanderson K, Corry J, Lapsley H. Utilising survey data to inform public policy: comparison of the cost-effectiveness of treatment of ten mental disorders. Br J Psychiatry. 2004 Jun;184:526-33. doi: 10.1192/bjp.184.6.526. PMID 15172947
- [Background] Kaltenthaler E, Parry G, Beverley C, Ferriter M. Computerised cognitive-behavioural therapy for depression: systematic review. Br J Psychiatry. 2008 Sep;193(3):181-4. doi: 10.1192/bjp.bp.106.025981. PMID 18757972
- [Background] Marks I, Cavanagh K. Computer-aided psychological treatments: evolving issues. Annu Rev Clin Psychol. 2009;5:121-41. doi: 10.1146/annurev.clinpsy.032408.153538. PMID 19327027
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Cuijpers P, Marks IM, van Straten A, Cavanagh K, Gega L, Andersson G. Computer-aided psychotherapy for anxiety disorders: a meta-analytic review. Cogn Behav Ther. 2009;38(2):66-82. doi: 10.1080/16506070802694776. PMID 20183688
- [Background] Titov N. Status of computerized cognitive behavioural therapy for adults. Aust N Z J Psychiatry. 2007 Feb;41(2):95-114. doi: 10.1080/00048670601109873. PMID 17464688
- [Background] Bender JL, Radhakrishnan A, Diorio C, Englesakis M, Jadad AR. Can pain be managed through the Internet? A systematic review of randomized controlled trials. Pain. 2011 Aug;152(8):1740-1750. doi: 10.1016/j.pain.2011.02.012. Epub 2011 May 11. PMID 21565446
- [Background] McCrone P, Knapp M, Proudfoot J, Ryden C, Cavanagh K, Shapiro DA, Ilson S, Gray JA, Goldberg D, Mann A, Marks I, Everitt B, Tylee A. Cost-effectiveness of computerised cognitive-behavioural therapy for anxiety and depression in primary care: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:55-62. doi: 10.1192/bjp.185.1.55. PMID 15231556
- [Background] McCrone P, Marks IM, Mataix-Cols D, Kenwright M, McDonough M. Computer-aided self-exposure therapy for phobia/panic disorder: a pilot economic evaluation. Cogn Behav Ther. 2009;38(2):91-9. doi: 10.1080/16506070802561074. PMID 19306148
- [Background] Hollinghurst S, Peters TJ, Kaur S, Wiles N, Lewis G, Kessler D. Cost-effectiveness of therapist-delivered online cognitive-behavioural therapy for depression: randomised controlled trial. Br J Psychiatry. 2010 Oct;197(4):297-304. doi: 10.1192/bjp.bp.109.073080. PMID 20884953
- [Background] Gerhards SA, de Graaf LE, Jacobs LE, Severens JL, Huibers MJ, Arntz A, Riper H, Widdershoven G, Metsemakers JF, Evers SM. Economic evaluation of online computerised cognitive-behavioural therapy without support for depression in primary care: randomised trial. Br J Psychiatry. 2010 Apr;196(4):310-8. doi: 10.1192/bjp.bp.109.065748. PMID 20357309
- [Background] Learmonth D, Rai S. Taking computerized CBT beyond primary care. Br J Clin Psychol. 2008 Mar;47(Pt 1):111-8. doi: 10.1348/014466507X248599. PMID 17939879
- [Background] Purves DG, Bennett M, Wellman N. An open trial in the NHS of Blues Begone: a new home based computerized CBT program. Behav Cogn Psychother. 2009 Oct;37(5):541-51. doi: 10.1017/S1352465809990282. Epub 2009 Aug 25. PMID 19703330
- [Background] Cavanagh K, Shapiro DA, Van Den Berg S, Swain S, Barkham M, Proudfoot J. The effectiveness of computerized cognitive behavioural therapy in routine care. Br J Clin Psychol. 2006 Nov;45(Pt 4):499-514. doi: 10.1348/014466505X84782. PMID 17076960
- [Background] Haby MM, Donnelly M, Corry J, Vos T. Cognitive behavioural therapy for depression, panic disorder and generalized anxiety disorder: a meta-regression of factors that may predict outcome. Aust N Z J Psychiatry. 2006 Jan;40(1):9-19. doi: 10.1080/j.1440-1614.2006.01736.x. PMID 16403033
- [Background] Gellatly J, Bower P, Hennessy S, Richards D, Gilbody S, Lovell K. What makes self-help interventions effective in the management of depressive symptoms? Meta-analysis and meta-regression. Psychol Med. 2007 Sep;37(9):1217-28. doi: 10.1017/S0033291707000062. Epub 2007 Feb 19. PMID 17306044
- [Background] Warmerdam L, van Straten A, Twisk J, Riper H, Cuijpers P. Internet-based treatment for adults with depressive symptoms: randomized controlled trial. J Med Internet Res. 2008 Nov 20;10(4):e44. doi: 10.2196/jmir.1094. PMID 19033149
- [Background] de Graaf LE, Gerhards SA, Arntz A, Riper H, Metsemakers JF, Evers SM, Severens JL, Widdershoven G, Huibers MJ. Clinical effectiveness of online computerised cognitive-behavioural therapy without support for depression in primary care: randomised trial. Br J Psychiatry. 2009 Jul;195(1):73-80. doi: 10.1192/bjp.bp.108.054429. PMID 19567900
- [Background] Waller R, Gilbody S. Barriers to the uptake of computerized cognitive behavioural therapy: a systematic review of the quantitative and qualitative evidence. Psychol Med. 2009 May;39(5):705-12. doi: 10.1017/S0033291708004224. Epub 2008 Sep 24. PMID 18812006
- [Background] Kaltenthaler E, Sutcliffe P, Parry G, Beverley C, Rees A, Ferriter M. The acceptability to patients of computerized cognitive behaviour therapy for depression: a systematic review. Psychol Med. 2008 Nov;38(11):1521-30. doi: 10.1017/S0033291707002607. Epub 2008 Jan 21. PMID 18205964
- [Background] Wangberg SC, Gammon D, Spitznogle K. In the eyes of the beholder: exploring psychologists' attitudes towards and use of e-therapy in Norway. Cyberpsychol Behav. 2007 Jun;10(3):418-23. doi: 10.1089/cpb.2006.9937. PMID 17594266
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Proudfoot J, Ryden C, Everitt B, Shapiro DA, Goldberg D, Mann A, Tylee A, Marks I, Gray JA. Clinical efficacy of computerised cognitive-behavioural therapy for anxiety and depression in primary care: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:46-54. doi: 10.1192/bjp.185.1.46. PMID 15231555
- [Background] Bellon JA, Moreno-Kustner B, Torres-Gonzalez F, Monton-Franco C, GildeGomez-Barragan MJ, Sanchez-Celaya M, Diaz-Barreiros MA, Vicens C, de Dios Luna J, Cervilla JA, Gutierrez B, Martinez-Canavate MT, Olivan-Blazquez B, Vazquez-Medrano A, Sanchez-Artiaga MS, March S, Motrico E, Ruiz-Garcia VM, Brangier-Wainberg PR, Del Mar Munoz-Garcia M, Nazareth I, King M; predictD group. Predicting the onset and persistence of episodes of depression in primary health care. The predictD-Spain study: methodology. BMC Public Health. 2008 Jul 25;8:256. doi: 10.1186/1471-2458-8-256. PMID 18657275
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Background] Norman SB, Cissell SH, Means-Christensen AJ, Stein MB. Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety. 2006;23(4):245-9. doi: 10.1002/da.20182. PMID 16688739
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] van Hout BA, Al MJ, Gordon GS, Rutten FF. Costs, effects and C/E-ratios alongside a clinical trial. Health Econ. 1994 Sep-Oct;3(5):309-19. doi: 10.1002/hec.4730030505. PMID 7827647
- [Background] Fenwick E, Claxton K, Sculpher M. Representing uncertainty: the role of cost-effectiveness acceptability curves. Health Econ. 2001 Dec;10(8):779-87. doi: 10.1002/hec.635. PMID 11747057
- [Background] Fenwick E, Byford S. A guide to cost-effectiveness acceptability curves. Br J Psychiatry. 2005 Aug;187:106-8. doi: 10.1192/bjp.187.2.106. PMID 16055820
- [Derived] Barcelo-Soler A, Garcia-Campayo J, Araya R, Doukani A, Gili M, Garcia-Palacios A, Mayoral F, Montero-Marin J. Working alliance in low-intensity internet-based cognitive behavioral therapy for depression in primary care in Spain: A qualitative study. Front Psychol. 2023 Mar 29;14:1024966. doi: 10.3389/fpsyg.2023.1024966. eCollection 2023. PMID 37063543
- [Derived] Mira A, Soler C, Alda M, Banos R, Castilla D, Castro A, Garcia-Campayo J, Garcia-Palacios A, Gili M, Hurtado M, Mayoral F, Montero-Marin J, Botella C. Exploring the Relationship Between the Acceptability of an Internet-Based Intervention for Depression in Primary Care and Clinical Outcomes: Secondary Analysis of a Randomized Controlled Trial. Front Psychiatry. 2019 May 10;10:325. doi: 10.3389/fpsyt.2019.00325. eCollection 2019. PMID 31133899
- [Derived] Romero-Sanchiz P, Nogueira-Arjona R, Garcia-Ruiz A, Luciano JV, Garcia Campayo J, Gili M, Botella C, Banos R, Castro A, Lopez-Del-Hoyo Y, Perez Ara MA, Modrego-Alarcon M, Mayoral Cleries F. Economic evaluation of a guided and unguided internet-based CBT intervention for major depression: Results from a multi-center, three-armed randomized controlled trial conducted in primary care. PLoS One. 2017 Feb 27;12(2):e0172741. doi: 10.1371/journal.pone.0172741. eCollection 2017. PMID 28241025
- [Derived] Montero-Marin J, Araya R, Perez-Yus MC, Mayoral F, Gili M, Botella C, Banos R, Castro A, Romero-Sanchiz P, Lopez-Del-Hoyo Y, Nogueira-Arjona R, Vives M, Riera A, Garcia-Campayo J. An Internet-Based Intervention for Depression in Primary Care in Spain: A Randomized Controlled Trial. J Med Internet Res. 2016 Aug 26;18(8):e231. doi: 10.2196/jmir.5695. PMID 27565118
- [Derived] Lopez-del-Hoyo Y, Olivan B, Luciano JV, Mayoral F, Roca M, Gili M, Andres E, Serrano-Blanco A, Collazo F, Araya R, Banos R, Botella C, Magallon R, Garcia-Campayo J. Low intensity vs. self-guided internet-delivered psychotherapy for major depression: a multicenter, controlled, randomized study. BMC Psychiatry. 2013 Jan 11;13:21. doi: 10.1186/1471-244X-13-21. PMID 23312003
- See also: Official website of the Spanish Research Network in Primary Care (Rediapp) — http://www.rediapp.org/